CLINICAL TRIAL: NCT00491985
Title: Safety and Immunogenicity of 2 Formulations of an Intramuscular A/H5N1 Pandemic Influenza Vaccine in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GPA04
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Influenza; Orthomyxoviridae Infections; Influenza A Virus Infection
Keywords: Influenza A/H5N1 Virus; Influenza Pandemic; Orthomyxoviridae Infections
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections

ARMS (3):
- Study Group 1 (Experimental): Subjects aged 9 to 17 years
  Interventions: Biological: A/H5N1 Inactivated, split-virion pandemic influenza vaccine
- Study Group 2 (Experimental): Subjects aged 3 to 8 years
  Interventions: Biological: A/H5N1 Inactivated, split virion pandemic influenza vaccine
- Study Group 3 (Experimental): Subjects aged 6 to 35 months
  Interventions: Biological: A/H5N1 Inactivated, split virion pandemic influenza vaccine

INTERVENTIONS:
Biological: A/H5N1 Inactivated, split-virion pandemic influenza vaccine — 0.5 mL, Intramuscular
  Arms: Study Group 1
Biological: A/H5N1 Inactivated, split virion pandemic influenza vaccine — 0.5 mL, Intramuscular
  Arms: Study Group 2
Biological: A/H5N1 Inactivated, split virion pandemic influenza vaccine — 0.25 mL, Intramuscular
  Arms: Study Group 3

SUMMARY:
This is an open, randomized, multicenter clinical trial.

Objectives:

* To describe the safety profiles during the 21 days following each primary and booster injection.
* To describe the immune response 21 days after each primary and booster injection of each formulation.
* To describe the antibody persistence after the first vaccination

ELIGIBILITY:
Inclusion Criteria :

All subjects:

* Able to attend all scheduled visits and to comply with all trial procedures.

Children/Adolescents aged ≥ 2 years to < 18 years:

* Aged ≥ 2 years to < 18 years on the day of inclusion.
* Informed Consent Form signed by one parent or another legal representative and by an independent witness if the parent/legal representative is illiterate.
* For a female, inability to bear a child or negative urine pregnancy test (as applicable).
* For a female of child-bearing potential, use of an effective method of contraception or abstinence for at least 4 weeks prior to the first vaccination and at least 4 weeks after the last vaccination (as applicable).

Infants/toddlers aged ≥ 6 months to < 2 years:

* Aged ≥ 6 months to < 2 years on the day of inclusion.
* Born at full term of pregnancy (≥ 37 weeks) with a birth weight ≥ 2 kg.
* Informed Consent Form signed by one parent/legally acceptable representative and an independent witness if the parent/legally acceptable representative is illiterate.
* Subject who completed vaccination according to the national immunization schedule.

Exclusion Criteria :

All subjects:

* Participation in another clinical trial in the 4 weeks preceding the first trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroid therapy.
* Systemic hypersensitivity to any of the vaccine components or history of life threatening reaction to the trial vaccine or a vaccine containing the same substances (egg proteins, chick proteins, thimerosal, aluminum, neomycin, formaldehyde, and octoxinol 9).
* Chronic illness at a stage that could interfere with trial conduct or completion.
* Blood or blood-derived products received in the past 3 months.
* Any vaccination in the 4 weeks preceding the first trial vaccination.
* Vaccination planned in the 4 weeks following any trial vaccination.
* History of the H5N1 infection (confirmed either clinically, serologically or virologically).
* Known HIV, Hepatitis B (HBsAg) or Hepatitis C seropositivity.
* Previous vaccination with an avian flu vaccine.
* Subject at high risk of the H5N1 infection during the trial.
* Thrombocytopenia or bleeding disorder contraindicating IM vaccination.
* Febrile illness (rectal equivalent temperature ≥ 38.0°C) on the day of inclusion.

Children/Adolescents aged ≥ 2 years to < 18 years:

* Breast-feeding mothers.
* Current alcohol abuse or drug addiction that may interfere with the subject's ability to comply with trial procedures (if applicable, depending on the subject's age).

Infants/toddlers aged ≥ 6 months to < 2 years:

* History of seizures.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 240 (Actual)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To describe safety following administration of A/H5N1 inactivated split virion pandemic influenza vaccine. | 21 Days post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc
Locations (1):
- Bangkok, Thailand

REFERENCES:
- [Derived] Chotpitayasunondh T, Thisyakorn U, Pancharoen C, Pepin S, Nougarede N. Safety, humoral and cell mediated immune responses to two formulations of an inactivated, split-virion influenza A/H5N1 vaccine in children. PLoS One. 2008;3(12):e4028. doi: 10.1371/journal.pone.0004028. Epub 2008 Dec 29. PMID 19112513
- See also: Related Info — http://www.sanofipasteur.com